CLINICAL TRIAL: NCT03772964
Title: A Pilot Study: Metformin as an Inflammatory Modulating Therapy in Older Adults Without Diabetes
Brief Title: Effects of Metformin in a Non-Diabetic Patient Population
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brian Zuckerbraun (Other)
Responsible Party: Sponsor-Investigator, Brian Zuckerbraun, Chief, Division of General/Trauma and Acute Care Surgery, Professor of Surgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PRO17100535
Record Dates: First submitted 2018-02-28; First posted 2018-12-12 (Actual); Results first posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Inflammatory Response
Keywords: prefrail; non-diabetic; metformin; thrombosis; microbiome; cellular respiration; short physical performance batter
MeSH Terms: conditions — Thrombosis | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Subjects will act as their own controls: data will be collect on each subject at baseline, throughout exposure and following, exposure to metformin.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 500mg exposure (Experimental): Subjects will be exposed to 500mg of daily MetFORMIN Hydrochloride ER for up to 90 days.
  Interventions: Drug: MetFORMIN Hydrochloride ER
- 1000mg exposure (Experimental): Subjects will be exposed to 1000mg of daily MetFORMIN Hydrochloride ER for up to 90 days.
  Interventions: Drug: MetFORMIN Hydrochloride ER
- 1500mg exposure (Experimental): Subjects will be exposed to 1500mg of daily MetFORMIN Hydrochloride ER for up to 90 days.
  Interventions: Drug: MetFORMIN Hydrochloride ER
- Placebo (Placebo Comparator): Subjects will be exposed to placebo for up to 90 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MetFORMIN Hydrochloride ER — Subjects will be exposed to 500mg, 1000mg, or 1500mg of daily ER Metformin, by mouth, for up to 90 days. Subjects will have their venous blood sampled and baseline, throughout the trial, and following completion of their metformin exposure.
  Other Names: Metformin ER
  Arms: 1000mg exposure; 1500mg exposure; 500mg exposure
Drug: Placebo — Subjects will be exposed to placebo, by mouth, for up to 90 days. Subjects will have their venous blood sampled and baseline, throughout the trial, and following completion of their metformin exposure.
  Arms: Placebo

SUMMARY:
Metformin has a well-established safety profile and it has become clear that metformin has additional salutary effects, including anti-inflammatory, anti-aging, and anti-thrombotic properties. In this study, subjects will provide both venous blood samples and stool samples in addition to completing cognitive and physiologic testing at baseline, throughout a 90 day exposure to metformin, and 30 days following exposure to metformin in order to evaluate their immune, microbiome, cellular respiration, thrombotic, and inflammatory responses.

DETAILED DESCRIPTION:
Metformin is considered first-line therapy for patients with type two diabetes with hyperglycemia that cannot be controlled with lifestyle alone. Unlike other oral medications, metformin is favored for its insulin-sensitizing effects resulting in improved glycemic control, weight loss, and overall improvement of metabolic syndrome. Over the past fifteen years, metformin has received significant attention for its other potential therapeutic uses. Metformin has been found to decrease the rate of age-related illness progression improving longevity, especially in the setting of cancer. Recent clinical trials across multiple disease states have shown metformin to decrease all-cause mortality in diabetic and non-diabetic patients. Additionally, in both animal models and human trails, metformin has been shown to decrease the risk of arterial and venous thrombosis without affecting bleeding time through its interaction with platelet mitochondria. Although the mechanisms by which metformin effects longevity is an active area of both basic science and clinical research, it clearly has anti-inflammatory properties which are both independent and dependent of glycemic control. Recently, surgical outcomes have focused on optimizing older, deconditioned patients prior to the operation with varying protocols referred to as prehabilitation. These programs work to improve the body's response to the surgical stress resulting in improved wound healing, decreased postoperative complications, and decreased hospital length of stay. The affect of metformin, like increasing physical activity, has widespread affects on physiology. The investigators, therefore, hypothesize that metformin administration to non-diabetic adults will improve clinical outcomes to physiologic stress by improving underlying immune and inflammatory responses, that can be deleterious.

Subjects will have venous samples collected to better understand the cellular response to inflammation, thrombosis, and cellular respiration at baseline, at 4 time points throughout the 90 day exposure to metformin, and 30 days following the completion of exposure to metformin. At the same time points, subjects will have stool samples collected in order to assess changes in their microbiome. Finally, subjects will undergo cognitive testing through the NIH toolbox as well as physiologic testing including (six-minute walk test, grip strength as measured by a dynamometer, and a short physical performance battery) at baseline, after 90 days of exposure, and again 30 days after the completion of exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥55 and ≤85 years of age
2. Non-diabetic
3. Adjusted risk analysis index (RAI) 20-42
4. Estimated glomerular filtration rate >45
5. No evidence of hepatic dysfunction on comprehensive metabolic panel
6. No clinical evidence of cardiac failure
7. Existing University of Pittsburgh Medical Center Patients

Exclusion Criteria:

1. Hypersensitivity to metformin or any component of the formulation
2. Acute or chronic metabolic acidosis with or without coma
3. Pregnant or breastfeeding females
4. Evidence or history of hepatic, renal, or cardiopulmonary failure
5. Excessive acute or chronic ethanol use
6. Planned or known hospital admission, exposure to anesthesia, or surgical intervention 30 days prior to study or scheduled 30 days after the trial initiation
7. Laboratory analysis showing HbgA1c >6.1 or eGFR <44 on baseline labs

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Zuckerbraun, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no current plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Randriamboavonjy V, Mann WA, Elgheznawy A, Popp R, Rogowski P, Dornauf I, Drose S, Fleming I. Metformin reduces hyper-reactivity of platelets from patients with polycystic ovary syndrome by improving mitochondrial integrity. Thromb Haemost. 2015 Aug 31;114(3):569-78. doi: 10.1160/TH14-09-0797. Epub 2015 May 21. PMID 25993908
- [Background] Xin G, Wei Z, Ji C, Zheng H, Gu J, Ma L, Huang W, Morris-Natschke SL, Yeh JL, Zhang R, Qin C, Wen L, Xing Z, Cao Y, Xia Q, Lu Y, Li K, Niu H, Lee KH, Huang W. Metformin Uniquely Prevents Thrombosis by Inhibiting Platelet Activation and mtDNA Release. Sci Rep. 2016 Nov 2;6:36222. doi: 10.1038/srep36222. PMID 27805009
- [Background] Alazawi W, Pirmadjid N, Lahiri R, Bhattacharya S. Inflammatory and Immune Responses to Surgery and Their Clinical Impact. Ann Surg. 2016 Jul;264(1):73-80. doi: 10.1097/SLA.0000000000001691. PMID 27275778
- [Background] Kato M, Suzuki H, Murakami M, Akama M, Matsukawa S, Hashimoto Y. Elevated plasma levels of interleukin-6, interleukin-8, and granulocyte colony-stimulating factor during and after major abdominal surgery. J Clin Anesth. 1997 Jun;9(4):293-8. doi: 10.1016/s0952-8180(97)00006-8. PMID 9195352
- [Background] Lin E, Calvano SE, Lowry SF. Inflammatory cytokines and cell response in surgery. Surgery. 2000 Feb;127(2):117-26. doi: 10.1067/msy.2000.101584. PMID 10686974
- [Background] Jansson K, Redler B, Truedsson L, Magnuson A, Matthiessen P, Andersson M, Norgren L. Intraperitoneal cytokine response after major surgery: higher postoperative intraperitoneal versus systemic cytokine levels suggest the gastrointestinal tract as the major source of the postoperative inflammatory reaction. Am J Surg. 2004 Mar;187(3):372-7. doi: 10.1016/j.amjsurg.2003.12.019. PMID 15006565
- [Background] Whelan SP, Zuckerbraun BS. Mitochondrial signaling: forwards, backwards, and in between. Oxid Med Cell Longev. 2013;2013:351613. doi: 10.1155/2013/351613. Epub 2013 May 29. PMID 23819011
- [Background] Waltz P, Carchman EH, Young AC, Rao J, Rosengart MR, Kaczorowski D, Zuckerbraun BS. Lipopolysaccaride induces autophagic signaling in macrophages via a TLR4, heme oxygenase-1 dependent pathway. Autophagy. 2011 Mar;7(3):315-20. doi: 10.4161/auto.7.3.14044. PMID 21307647
- [Background] Keel M, Schregenberger N, Steckholzer U, Ungethum U, Kenney J, Trentz O, Ertel W. Endotoxin tolerance after severe injury and its regulatory mechanisms. J Trauma. 1996 Sep;41(3):430-7; discussion 437-8. doi: 10.1097/00005373-199609000-00008. PMID 8810959
- [Background] Loomba R, Lutchman G, Kleiner DE, Ricks M, Feld JJ, Borg BB, Modi A, Nagabhyru P, Sumner AE, Liang TJ, Hoofnagle JH. Clinical trial: pilot study of metformin for the treatment of non-alcoholic steatohepatitis. Aliment Pharmacol Ther. 2009 Jan;29(2):172-82. doi: 10.1111/j.1365-2036.2008.03869.x. Epub 2008 Oct 9. PMID 18945255
- [Background] Hou X, Song J, Li XN, Zhang L, Wang X, Chen L, Shen YH. Metformin reduces intracellular reactive oxygen species levels by upregulating expression of the antioxidant thioredoxin via the AMPK-FOXO3 pathway. Biochem Biophys Res Commun. 2010 May 28;396(2):199-205. doi: 10.1016/j.bbrc.2010.04.017. Epub 2010 Apr 14. PMID 20398632
- [Background] Harrison DE, Strong R, Sharp ZD, Nelson JF, Astle CM, Flurkey K, Nadon NL, Wilkinson JE, Frenkel K, Carter CS, Pahor M, Javors MA, Fernandez E, Miller RA. Rapamycin fed late in life extends lifespan in genetically heterogeneous mice. Nature. 2009 Jul 16;460(7253):392-5. doi: 10.1038/nature08221. Epub 2009 Jul 8. PMID 19587680
- [Background] Algire C, Moiseeva O, Deschenes-Simard X, Amrein L, Petruccelli L, Birman E, Viollet B, Ferbeyre G, Pollak MN. Metformin reduces endogenous reactive oxygen species and associated DNA damage. Cancer Prev Res (Phila). 2012 Apr;5(4):536-43. doi: 10.1158/1940-6207.CAPR-11-0536. Epub 2012 Jan 18. PMID 22262811
- [Background] Smith DL Jr, Elam CF Jr, Mattison JA, Lane MA, Roth GS, Ingram DK, Allison DB. Metformin supplementation and life span in Fischer-344 rats. J Gerontol A Biol Sci Med Sci. 2010 May;65(5):468-74. doi: 10.1093/gerona/glq033. Epub 2010 Mar 19. PMID 20304770
- [Background] Pernicova I, Korbonits M. Metformin--mode of action and clinical implications for diabetes and cancer. Nat Rev Endocrinol. 2014 Mar;10(3):143-56. doi: 10.1038/nrendo.2013.256. Epub 2014 Jan 7. PMID 24393785

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 500mg Exposure | 1000mg Exposure | 1500mg Exposure | Placebo
Started | 8 | 8 | 8 | 8
Completed | 7 (Could not attend final in-person evaluation due to COVID-19 shut down limitations) | 8 | 8 | 8
Not Completed | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 500mg Exposure | 1000mg Exposure | 1500mg Exposure | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (6) | 70 (6) | 71 (4) | 68 (6) | 70 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 4 | 5 | 17
  Male | 3 | 5 | 4 | 3 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 0 | 3
  White | 7 | 7 | 7 | 8 | 29
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Ex Vivo Cytokine Response of Peripheral Blood Mononucleocytes (PBMC) to Inflammatory Stimuli Compared to Baseline, Throughout Exposure, and Following Exposure to Metformin.
Description: Venous blood samples will be gathered throughout the study in order to quantify the changes in cytokine expression (FN-γ, IL-10, IL12p40, IL-12p70, IL-1α, IL1β, IL-2, IL-6, IL-8, IP-10, MCP-1, MIP-1α, MIP-1β, TNF-α) following ex vivo PBMC exposure to endotoxin.
Time Frame: Day 0 (baseline), 30, 60, 90, and 120 (30 days post metformin exposure)
Population: Samples collected. Results were not yielded as they were not adequate to run samples with the available staffing.
Arm/Group | 500mg Exposure | 1000mg Exposure | 1500mg Exposure | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Quantify the Bacterial Population Profile of the Microbiome Via Stool Samples.
Description: Bacterial communities using 16S rRNA sequencing in relationship to metformin dosing over time. Species richness or diversity in the sample is measured by Choa1 metric. Chao1 is an estimate of how many species are present in an ecosystem. In general, having more species is considered to be "healthier" and these values typically range from 100-200 for fecal samples. The Chao1 index over numerous samples across time are explored to understand treatment effects.
Time Frame: Day 0 (baseline), 30, 60, 90, and 120 (30 days post metformin exposure)
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | 500mg Exposure | 1000mg Exposure | 1500mg Exposure | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8
Index
  Day 0 | 136.5 (19.0) | 107.6 (13.3) | 128.1 (10.5) | 141.5 (15)
  Day 30 | 139.9 (16.2) | 130.7 (19.4) | 128.1 (13.2) | 144.75 (13.2)
  Day 60 | 121.4 (20.8) | 137.9 (17.7) | 128.6 (12.7) | 134.3 (9.8)
  Day 90 | 137.8 (27.8) | 135 (18.9) | 138.2 (10.3) | 152 (20.5)
  Day 120 | 134 (23.6) | 142.2 (17.3) | 144.2 (16.5) | 159.2 (5.7)
Statistical Analysis 1: Comparison: 500mg Exposure vs 1000mg Exposure vs 1500mg Exposure vs Placebo; Beta Diversity - Differences between Samples and Sample groups; Test type: Superiority — Comparisons between samples and sample groups (beta-diversity), were evaluated with ADONIS (aka PERMANOVA) comparisons of differences between sample groups; p < 0.01, ADONISBeta Diversity; Comparisons between samples and sample groups (beta-diversity) were evaluated with ADONIS (aka PERMANOVA); R2 = 0.071435 — R2 values estimate the amount of variation explained by each variable

3. Secondary Outcome: Measure the Rate of Clotting of Peripheral Blood With Whole Blood Aggregometry in Response to Collagen.
Description: Aggregometry area under the curve with the Y-axis being % aggregometry and the X-axis time in minutes.
Time Frame: Day 0 (baseline), 30, 60, 90, and 120 (30 days post metformin exposure)
Population: Samples were collected and processed at each time point for each participant. When sample processing did not yeild any result (processing failure) no data could be yeilded and therefore can not be presented.
Measure: Mean (Standard Deviation); unit: arbitrary units*mins
Arm/Group | 500mg Exposure | 1000mg Exposure | 1500mg Exposure | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8
arbitrary units*mins
  0 days | 56.3 (40) | 67 (38) | 196 (376) | 83.3 (69)
  30 day change from day 0 | -34.7 (24.5) | 8.9 (50.1) | -166.7 (409) | -29.6 (104.8)
  60 days change from day 0 | -28.3 (54) | -23.5 (44.5) | -139.8 (376.3) | -49.4 (86.7)
  90 days change from day 0: number analyzed (Participants) | 6 | 5 | 7 | 5
  90 days change from day 0 | 1.6 (57.6) | 2.4 (84.5) | -222.5 (456.2) | -66.6 (102.6)
  120 days change from day 0: number analyzed (Participants) | 6 | 4 | 6 | 6
  120 days change from day 0 | -49.2 (84.2) | 1.0 (28.9) | -196.7 (410.6) | -47.6 (103.0)
Statistical Analysis 1: Comparison: 500mg Exposure vs 1000mg Exposure vs 1500mg Exposure vs Placebo; Test type: Superiority; p = 0.6057, ANOVA

4. Secondary Outcome: Measure the Rate of Thrombosis of Peripheral Blood.
Description: The endpoints for isolated platelets include platelet activation as measured by FACS for CD62p.
Time Frame: Day 0 (baseline), 30, 60, 90, and 120 (30 days post metformin exposure)
Population: These data were not able to be collected due to storage issues and lab shutdowns during the COVID-19 pandemic.
Arm/Group | 500mg Exposure | 1000mg Exposure | 1500mg Exposure | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Changes From Baseline in Short Physical Performance Battery (SPPB) During and Following Exposure to Metformin.
Description: The SPPB is a group of measures that combines the results of the gait speed, chair stand and balance tests. The minimum is zero (worse performance) and the maximum is 12 (best performance).
Time Frame: Day 0 (baseline), 90, and 120 (30 days post metformin exposure)
Population: Notably, one patient in the 500mg and 1000mg group was unable to finish the 120d testing secondary to COVID-19 limitations.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Placebo: Participants were exposed to oral placebo for up to 90 days.
Arm/Group | 500mg Exposure | 1000mg Exposure | 1500mg Exposure | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8
Units on a scale
  0d | 11.2 (.9) | 10.8 (1.3) | 11.1 (0.9) | 10.6 (1.3)
  90d, change from 0d | -0.3 (1.4) | 0.4 (0.7) | 0.4 (0.5) | 1.0 (1.0)
  120d, change from 0d: number analyzed (Participants) | 7 | 7 | 8 | 8
  120d, change from 0d | 0 (0.6) | 0.2 (1.0) | 0.3 (1.3) | 0.5 (.8)
Statistical Analysis 1: Comparison: 500mg Exposure vs 1000mg Exposure vs 1500mg Exposure vs Placebo; Test type: Superiority; p < 0.001, ANOVA

6. Secondary Outcome: Changes From Baseline in Grip Strength Via a Dynamometer During and Following Exposure to Metformin.
Description: Grip strength over time.
Time Frame: Day 0 (baseline), 90, and 120 (30 days post metformin exposure)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Placebo: Subjects exposed to placebo for up to 90d
Arm/Group | 500mg Exposure | 1000mg Exposure | 1500mg Exposure | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8
mmHg
  0 days | 28.2 (10.3) | 28.9 (8.3) | 25.7 (7.8) | 25.7 (9.2)
  90 days, compared to 0 days | -5.3 (12.5) | -0.4 (3.1) | -.2 (2.1) | -.3 (3.5)
  120 days, compared to 0 days: number analyzed (Participants) | 7 | 7 | 8 | 8
  120 days, compared to 0 days | .1 (4.8) | 1.1 (2.7) | .3 (3.0) | -.6 (2.0)
Statistical Analysis 1: Comparison: 500mg Exposure vs 1000mg Exposure vs 1500mg Exposure vs Placebo; Test type: Superiority; p = 0.69, ANOVA

7. Secondary Outcome: Mitochondrial Respiration in Both PBMCs and Platelets.
Description: Oxidative phosphorylation, respiration, and complex activity will be tested using an Oroboros respirometer.
Time Frame: Day 0 (baseline), 30, 60, 90, and 120 (30 days post metformin exposure)
Population: Samples were collected. Cell processing did not allow for the analysis of any data from collected samples. No data were therefore able to be collected.
Arm/Group | 500mg Exposure | 1000mg Exposure | 1500mg Exposure | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Mitochondrial Content in Both PBMCs and Platelets.
Description: Mitochondrial content will be measured by staining for mitotracker, and mitochondrial DNA oxidation will be determined by co-localizing staining for 8-hydroxydeoxyguanosine (8-OHdG). Markers of autophagy will be determined by measuring LC-3 flux, p62, beclin-1, and ATG7 protein levels.
Time Frame: Day 0 (baseline), 30, 60, 90, and 120 (30 days post metformin exposure)
Population: as for outcome 7
Arm/Group | 500mg Exposure | 1000mg Exposure | 1500mg Exposure | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Measure Biogenesis of PBMCs.
Description: Biogenesis will be determined by measuring RNA for PGC1a, NRF-1, and Tfam.
Time Frame: Day 0 (baseline), 30, 60, 90, and 120 (30 days post metformin exposure)
Population: as for outcome 7
Arm/Group | 500mg Exposure | 1000mg Exposure | 1500mg Exposure | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the time of randomization for 120 days.
Description: Unexpected serious adverse events including significant illness, hospitalization, emergent or urgent surgery or procedure, psychiatric hospitalization or inpatient rehabilitation, would require the study team to discontinue the subject's participation.
Arm/Group | 500mg Exposure | 1000mg Exposure | 1500mg Exposure | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 5/8 | 3/8 | 6/8 | 5/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 500mg Exposure (N=8) | 1000mg Exposure (N=8) | 1500mg Exposure (N=8) | Placebo (N=8)
Gastrointestinal symptoms (Gastrointestinal disorders) | 5 (5) | 1 (1) | 4 (4) | 5 (5) — Bloating, flatus, nausea, heartburn, or diarrhea were captured as a single entity and summarized as gastrointestinal symptoms.
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) — Upper respiratory infection including sinusitis, common cold, congestion
Joint pain or fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2) — Joint pain or fracture

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT03772964/Prot_SAP_000.pdf